CLINICAL TRIAL: NCT03312374
Title: Circulating Tumor DNA as a Prognostic Marker for Postoperative Relapse in Early and Intermediate Stage Colorectal Cancer:A Prospective, Multicenter,Observational, Single-Blinded Controlled Study
Brief Title: ctDNA as a Prognostic Marker for Postoperative Relapse in Early and Intermediate Stage Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Fudan University (Other); Zhejiang University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Clinical Professor, Sun Yat-sen University
Other Study IDs: CTDNA-CRC
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — The fresh tumor tissues/biopsies of each patient will be collected during the surgical resection. The peripheral blood samples of each patient will be collected at the following time points: 1) prior to the surgical treatment; 2) 3-7 days after the surgical resection; 3) every three months(starting from 6 months) until disease progression (up to 24 months).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- stage II CRC: Patients with stage II colorectal cancer
- stage III CRC: Patients with stage III colorectal cancer

SUMMARY:
By monitoring the serum ctDNA mutational profile using NGS, the present clinical trial aims to elucidate the correlation between the postoperative ctDNA status and the prognosis of patients with early and intermediate-stage colorectal cancer, and explore the possibility of clinical utility of serum ctDNA as a clinical index to predict postoperative relapse.

DETAILED DESCRIPTION:
Colorectal cancer (CRC), as one of the common malignant tumors with high mobidity and mortality, is a major health threat in China.Surgical resection is the conventional treatment for early and intermediate stageCRC, however, it is not curative and postoperative recurrenceremains a clinical dilemma.Early detection of recurrence by serum tumor biomarkers and Computed Tomography (CT) during follow-up can improve the overall survival of patients with surgical resection. Nevertheless, thecurrently available tumor biomarkers have limited sensitivity and specificity, and CT is associated with radiation exposure. Therefore, there is a need for a more effective and feasible methodfor the prediction of postoperative recurrence.

Circulating tumor DNA (ctDNA) is tumor-derived fragmented DNA with an average size of 170bp, mixed with cell free DNA (cfDNA) of other sources in blood circulation. Although the mechanisms of its release have not been fully addressed, apoptosis and/or necrosis of tumor cells and serum exosome are considered as its main source, which makes it a genomic reservoir of different tumor clones. Also, as its half-life is up to hours, ctDNA is reflecting the most up-to-date status of tumor genome. Hence, it allows for noninvasive molecular characterization of tumors,which can be qualitative, quantitative and used for disease monitoring.

The possibility of that ctDNA could be used to detect micrometastatic disease in patients received surgical resection was suggested in several studies. UsingNext Generation Sequencing (NGS),Newman et al. have shown that the serum level of ctDNA was correlated withtumor progress and prognosis in NSCLC. Isaac et al. demonstrated the postoperativectDNA level was associated with breast cancer progression, and it was more sensitive compared to CT scan for predicting the early relapse. Tie et al. examined the postoperative ctDNA level of 1046 plasma samples from a prospective cohort of 230 patients with resected stage II CRC by NGS, and their results demonstrated that recurrence happened in 79% of the patients with positive postoperative ctDNA at median follow-up of 27 months, versus 9.8% in the negative postoperative ctDNA group.

By monitoring the serum ctDNA mutational profile using NGS, the present clinical trial aims to elucidate the correlation between the postoperative ctDNA status and the prognosis of patients with early and intermediate-stage colorectal cancer, and explore the possibility of clinical utility of serum ctDNA as a clinical index to predict postoperative relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age on the day of signing informed consent.
2. Patients must have histologically confirmed stage II/IIIcolorectal cancer.
3. Patients need to receive surgical resection.
4. Patients must have a performance status of ≤1 on the ECOG Performance Scale.
5. Patients must have survival of > 12 months after the index date
6. Written informed consent must be obtained from patient or patient's legal representative and ability for patient to comply with the requirements of the study.

Exclusion Criteria:

1. Patients received adjuvant treatment prior to the surgical resection.
2. Patients received blood transfusion two weeks before or during the surgical resection.
3. Patients who are positive for Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C.
4. Patients who are pregnant.
5. Patients who are alcoholic or drug abusers.
6. Patients with a history or current evidence of any condition or abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must have baseline evaluations performed prior to the study and must meet all inclusion and exclusion criteria. In addition, the patient must be thoroughly informed about all aspects of the study, including the study visit schedule and required evaluations and all regulatory requirements for informed consent. The written informed consent must be obtained from the patient prior to enrollment. The following criteria apply to all patients enrolled onto the study unless otherwise specified.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | through study completion, an average of 2 years
  The primary endpoint for this study is Disease Free Survival (DFS), which will be assessed using RECIST version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, MD.,PhD., Study Chair — Sun Yat-sen University
Locations (1):
- Medical Oncology,Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Guinney J, Dienstmann R, Wang X, de Reynies A, Schlicker A, Soneson C, Marisa L, Roepman P, Nyamundanda G, Angelino P, Bot BM, Morris JS, Simon IM, Gerster S, Fessler E, De Sousa E Melo F, Missiaglia E, Ramay H, Barras D, Homicsko K, Maru D, Manyam GC, Broom B, Boige V, Perez-Villamil B, Laderas T, Salazar R, Gray JW, Hanahan D, Tabernero J, Bernards R, Friend SH, Laurent-Puig P, Medema JP, Sadanandam A, Wessels L, Delorenzi M, Kopetz S, Vermeulen L, Tejpar S. The consensus molecular subtypes of colorectal cancer. Nat Med. 2015 Nov;21(11):1350-6. doi: 10.1038/nm.3967. Epub 2015 Oct 12. PMID 26457759
- [Result] Rolfo C, Castiglia M, Hong D, Alessandro R, Mertens I, Baggerman G, Zwaenepoel K, Gil-Bazo I, Passiglia F, Carreca AP, Taverna S, Vento R, Santini D, Peeters M, Russo A, Pauwels P. Liquid biopsies in lung cancer: the new ambrosia of researchers. Biochim Biophys Acta. 2014 Dec;1846(2):539-46. doi: 10.1016/j.bbcan.2014.10.001. Epub 2014 Oct 16. PMID 25444714
- [Result] Yu SC, Lee SW, Jiang P, Leung TY, Chan KC, Chiu RW, Lo YM. High-resolution profiling of fetal DNA clearance from maternal plasma by massively parallel sequencing. Clin Chem. 2013 Aug;59(8):1228-37. doi: 10.1373/clinchem.2013.203679. Epub 2013 Apr 19. PMID 23603797
- [Result] Newman AM, Bratman SV, To J, Wynne JF, Eclov NC, Modlin LA, Liu CL, Neal JW, Wakelee HA, Merritt RE, Shrager JB, Loo BW Jr, Alizadeh AA, Diehn M. An ultrasensitive method for quantitating circulating tumor DNA with broad patient coverage. Nat Med. 2014 May;20(5):548-54. doi: 10.1038/nm.3519. Epub 2014 Apr 6. PMID 24705333
- [Result] Garcia-Murillas I, Schiavon G, Weigelt B, Ng C, Hrebien S, Cutts RJ, Cheang M, Osin P, Nerurkar A, Kozarewa I, Garrido JA, Dowsett M, Reis-Filho JS, Smith IE, Turner NC. Mutation tracking in circulating tumor DNA predicts relapse in early breast cancer. Sci Transl Med. 2015 Aug 26;7(302):302ra133. doi: 10.1126/scitranslmed.aab0021. PMID 26311728
- [Result] Tie J, Wang Y, Tomasetti C, Li L, Springer S, Kinde I, Silliman N, Tacey M, Wong HL, Christie M, Kosmider S, Skinner I, Wong R, Steel M, Tran B, Desai J, Jones I, Haydon A, Hayes T, Price TJ, Strausberg RL, Diaz LA Jr, Papadopoulos N, Kinzler KW, Vogelstein B, Gibbs P. Circulating tumor DNA analysis detects minimal residual disease and predicts recurrence in patients with stage II colon cancer. Sci Transl Med. 2016 Jul 6;8(346):346ra92. doi: 10.1126/scitranslmed.aaf6219. PMID 27384348